CLINICAL TRIAL: NCT05949398
Title: Evaluation of the Prevalence and Type of Oral HPV Infection in Patients Who Are Positive to the PAP-test
Brief Title: Evaluation of the Prevalence of Oral HPV Infection in Patients Who Are Positive to the PAP-test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Principal Investigator, University of Catania
Other Study IDs: 121-27
Record Dates: First submitted 2023-06-24; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: HPV Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cytological sampling of oral mucosa cells in order to identify possible genetic material (DNA) of HPV. The tubes with the biological sample to be processed are labeled with the patient's master data. The material should be stored at +4°C or room temperature for no more than 3 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present cross-sectional study aims to assess the prevalence and type distribution of oral HPV infection in PAP-test-positive women aged ≥18 years. The means used in the present study will be the use of anamnestic questionnaires and exfoliative cytology tests at predetermined oral mucosal sites (lingual belly and dorsum, palate, and buccal mucosa).

DETAILED DESCRIPTION:
The present cross-sectional study aims to evaluate the prevalence and distribution of the type of oral HPV infection in PAP-test positive women.

aged ≥18 years. Sociodemographic and anamnestic data will be collected by questionnaire administration. Data collected will be age, marital status, number of sexual partners, HPV vaccination, oral sex, contraceptive use, systemic diseases, smoking, alcohol consumption, etc.. Next, patients will undergo oral cavity inspection and exfoliative cytology testing at predetermined oral mucosal sites (lingual belly and dorsum, palate, and buccal mucosa).

Sample taken sent for cytological analysis to determine the presence of viral DNAand possible typing.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with positive PAP test;
* Age ≥ 18 years

Exclusion Criteria:

* Female patients with negative PAP test
* Uncooperative patients
* Patients with mental deficits
* Age<18 years

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women older than 18 years of age who are PAP-test positive.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-13 (Estimated); Study Completion 2023-09-26 (Estimated)

PRIMARY OUTCOMES:
Prevalence and type of oral HPV infection in PAP-test positive patients | 1 Month
  Evaluation of the prevalence and type of oral HPV infection in PAP-test positive patients by objective examination of the oral cavity and performance of exfoliative cytology tests at oral mucosal sites predetermined (lingual belly and dorsum, palate, and buccal mucosa).
  The data will then be processed through the appropriate statistical examinations.
To assess whether there are any factors that may or may not promote the occurrence of oral HPV lesions in PAP-test positive patients, | 1 Month
  To assess whether there are any factors that may or may not promote the occurrence of oral HPV lesions in PAP-test positive patients, such as sociodemographic characteristics, diabetes, smoking, alcohol, HPV vaccination, etc. The data collected are as follows:
  * Collection of sociodemographic data by questionnaires (age, gender, civil status, education level, and occupation);
  * Collection of medical history data by questionnaires (smoking, alcohol consumption, diabetes or/and other systemic diseases, number of sexual partners, age of first intercourse, contraceptive use, type of contraceptive, HPV vaccination, sexual partners with genital/oral HPV infection).
  the following collected data will then be processed by statistical association surveys and uni and multivariate regression analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — University of Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Undecided